CLINICAL TRIAL: NCT00001120
Title: Oncogenic Viral Pathogenesis and Cancer Risk Factors Among Patients With the Acquired Immunodeficiency Syndrome: A Prospective Cohort Study
Brief Title: A Study of Patients With AIDS Syndrome
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Other Study IDs: ACTG A5035
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2008-09-12 (Estimated); Status verified 2006-05

CONDITIONS: Sarcoma, Kaposi; Lymphoma, Non-Hodgkin; HIV Infections; Lymphoma, AIDS-Related
Keywords: Prospective Studies; Sarcoma, Kaposi; Herpesvirus 4, Human; Acquired Immunodeficiency Syndrome; Cohort Studies; Risk Factors; Lymphoma, AIDS-Related; Antibodies, Viral; Lymphoproliferative Disorders; Viral Load; Herpesvirus, Kaposi Sarcoma-Associated; Translocation (Genetics)
MeSH Terms: conditions — Sarcoma, Kaposi; Lymphoma, Non-Hodgkin; HIV Infections; Lymphoma, AIDS-Related; Epstein-Barr Virus Infections; Acquired Immunodeficiency Syndrome; Lymphoproliferative Disorders; Translocation, Genetic

SUMMARY:
The purpose of this study is to find out why cancers develop in HIV-positive patients.

Cancer is a leading cause of death in AIDS patients. Common cancers in HIV-infected patients include Kaposi's sarcoma (KS) and non-Hodgkin's lymphoma (NHL), a cancer of the immune system. Risk factors include certain chemicals, viruses, and perhaps even anti-HIV drugs. Doctors would like to find out which risk factors are most important and how they relate to cancer in AIDS patients.

DETAILED DESCRIPTION:
AIDS-associated malignancy represents a model system for investigations of carcinogenesis. There are few human conditions in which cancer rates are of the magnitude they are in HIV infection. While studies have investigated pre-cancer markers in HIV-infected patients, they have not correlated these markers with tumor samples. This study contributes to understanding oncogenesis of HIV-associated malignancies by establishing a collection of tumors linked with pre-cancer sera and lymphocyte specimens, as well as prospective questionnaire data.

At study entry, patients receive a comprehensive physical exam. Clinic staff interview the patient to collect data regarding medication history (particularly antiretroviral exposure), diet, occupational history, substance abuse, and sexual practices. This information is used to identify behavioral and environmental factors contributing to oncogenesis. In addition, baseline blood samples are analyzed for HHV-8 and EBV levels, anti-EBV and anti-HHV-8 antibodies, CD23, Th2 cytokines, tumor growth factors, chromosomal translocations associated with NHL, and other potential predictors of malignancy. At Month 6 and annually thereafter, patient records are abstracted for data on vital status, AIDS-defining illnesses, medications, and most recent CD4+ T cell and HIV RNA levels. At Years 1, 2, and 3, patients undergo physical exams and blood tests for malignancy surveillance. Any malignancies are biopsied and analyzed for oncogene identification and virology. The medical records of patients who die on study are reviewed to determine the cause of death and to rule out unreported cancer. No treatment is provided by this study.

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this trial if you:

* Are HIV-positive.
* Have a CD4+ cell count of 200 cells/mm3 or below.
* Are 18 years of age or older.

Exclusion Criteria

You will not be eligible for this trial if you:

* Are not available for follow-up for at least 3 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5000

CONTACTS AND LOCATIONS:
Overall Officials: David A. Wohl, Study Chair — Univ of North Carolina; Ann C. Collier, Study Chair — Univ of Washington; William G. Powderly, Study Chair; Charles S. Rabkin, Principal Investigator
Locations (23):
- United States (23):
  - Willow Clinic, Menlo Park, California
  - San Francisco Gen Hosp, San Francisco, California
  - Marin County Specialty Clinic, San Rafael, California
  - San Mateo AIDS Program / Stanford Univ, Stanford, California
  - Stanford Univ Med Ctr, Stanford, California
  - Univ of Hawaii, Honolulu, Hawaii
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Charity Hosp / Tulane Univ Med School, New Orleans, Louisiana
  - Tulane Univ School of Medicine, New Orleans, Louisiana
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Harvard (Massachusetts Gen Hosp), Boston, Massachusetts
  - SUNY / Erie County Med Ctr at Buffalo, Buffalo, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Mem Sloan - Kettering Cancer Ctr, New York, New York
  - St Mary's Hosp (Univ of Rochester/Infectious Diseases), Rochester, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Duke Univ Med Ctr, Durham, North Carolina
  - Univ of Cincinnati, Cincinnati, Ohio
  - Case Western Reserve Univ, Cleveland, Ohio
  - MetroHealth Med Ctr, Cleveland, Ohio
  - Ohio State Univ Hosp Clinic, Columbus, Ohio
  - Univ of Washington, Seattle, Washington